CLINICAL TRIAL: NCT07229053
Title: Evaluation of the Factors Affecting the Length of Hospitalisation of Patients In Stroke Rehabilitation
Brief Title: Hospitalisation Duration in Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Naz Kalem, PM&R Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-1242
Record Dates: First submitted 2025-07-07; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Stroke Rehabilitation
Keywords: stroke rehabilitation; hospitalisation; inpatient rehabilitation duration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who stay hospital shorter than mean duration: The average length of hospital stay (weeks) of patients hospitalised due to hemiplegia since the opening of Etlik City Hospital will be determined. Patients will be divided into two groups as those hospitalised for shorter and longer than the average length of stay.
- patients who stay hospital longer than mean duration: The average length of hospital stay (weeks) of patients hospitalised due to hemiplegia since the opening of Etlik City Hospital will be determined. Patients will be divided into two groups as those hospitalised for shorter and longer than the average length of stay.

SUMMARY:
The stage at which functional recovery stops during the rehabilitation programme and which is one of the important determinants of the discharge decision is called "plateau". Although the definition of plateau is not clear, it is assessed with scales valid for a specific patient. Generally, plateau is not a stage in which functional recovery is completely terminated in stroke patients, but a period of pause. Detection of the plateau stage is important in planning the interruption of treatment and discharge of patients who continue inpatient rehabilitation programme. Factors causing plateau should be identified and necessary modifications should be made for effective continuation of the rehabilitation programme.The average length of hospital stay (weeks) of patients hospitalised due to hemiplegia since the opening of Etlik City Hospital will be determined. Patients will be divided into two groups as those hospitalised for shorter and longer than the average length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Followed by ischaemic or haemorrhagic stroke
* No more than 2 years have passed since the date of the incident
* Patients and their carers who are over 18 years of age

Exclusion Criteria:

* Cognitive or psychological impairment of the patient or carer
* The patient is discharged voluntarily or transferred to another department without completing the treatment
* Not volunteering to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who approved for inpatient stroke rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Scale | first day of inpatient rehabilitation, before discharged from hospital

SECONDARY OUTCOMES:
Berg Scale | first day of inpatient rehabilitation, before discharged from hospital
Mini Mental State Test | first day of inpatient rehabilitation
Beck Depression Scale | first day of inpatient rehabilitation
  Beck depression scale applied to patient
Beck depression scale | first day of inpatient rehabilitation
  beck depression scale applied to caregiver

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)